CLINICAL TRIAL: NCT03633721
Title: Acute Effects of Cannabis on Cognition and Mobility in Older HIV-infected and Uninfected Women
Brief Title: Acute Effects of Cannabis on Cognition and Mobility in Older HIV-infected and HIV-Un-infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018-9188; R21AG059505-01 (NIH)
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: HIV; AIDS; Aging
Keywords: mobility; cognition; WIHS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Participants will receive either cannabis or placebo on 1st visit and the opposite on the 2nd visit.
Who Masked: Participant, Care Provider
Masking Description: Neither participant nor care provider will be informed when cannabis/placebo are administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HIV positive; cannabis (Active Comparator): HIV positive women will be given cannabis and tested
  Interventions: Drug: Cannabis; Other: Placebo
- HIV positive; placebo (Placebo Comparator): HIV positive women will be given placebo and tested
  Interventions: Drug: Cannabis; Other: Placebo
- HIV negative; cannabis (Active Comparator): HIV negative women will be given cannabis and tested
  Interventions: Drug: Cannabis; Other: Placebo
- HIV negative; placebo (Placebo Comparator): HIV negative women will be given placebo and tested
  Interventions: Drug: Cannabis; Other: Placebo

INTERVENTIONS:
Drug: Cannabis — 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Other Names: Cannabis administered to HIV+ and HIV- women
Other: Placebo — 0% THC cigarettes will be administered to HIV negative women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Other Names: Placebo administered to HIV+ and HIV- women

SUMMARY:
The purpose of this study is to try to understand and explain why HIV-infected and uninfected women who use cannabis (marijuana) currently, or have used cannabis in the past, have higher risk of having experienced a fall in our earlier analyses in WIHS. This study will compare what happens when women are given cannabis compared with placebo, on measures of mobility, including walking speed under walking conditions that vary in terms of difficulty; for example normal walking and walking while reciting alternate letters of the alphabet, as well as measures of balance and cognition (for example attention, memory).

DETAILED DESCRIPTION:
Cannabis is the most prevalent drug used by adults aged 50 and older in the U.S., after alcohol and tobacco. Recent trends show dramatic increases in cannabis use among older U.S. adults, and rising cannabis tetrahydrocannabinol (THC) content. Cannabis intoxication acutely alters short-term memory, attention span, verbal fluency, reaction time, and psychomotor control. Heavy long term cannabis use has been associated with lasting impairments in verbal learning, memory, and attention that correlate with duration of use; however, other studies have found that cognitive deficits from cannabis are reversible and related to recent exposure. But studies on cannabis exposure and cognition are age limited by including only adolescents through middle-aged adults; effects of acute and long-term cannabis use on cognition among older adults are virtually unknown. Given the rising potency and increasing frequency of cannabis use among older adults, studies systematically examining the risks and benefits of cannabis use in older adults are urgently needed.

Cannabis use is particularly common in people living with HIV (PLWH), with 12- 56% prevalence rates compared to 9.5% in the general U.S. population. HIV has detrimental effects on both mobility and cognition, and similar to normal aging, mobility in patients with HIV may be influenced by cognitive function. Mild-to-moderate neurocognitive impairments (NCI), notably in attention and executive functions, remain highly prevalent and persist despite suppressive antiretroviral therapy, affecting almost half of PLWH. Little is known about the combined effects of cannabis use and HIV infection on cognition and mobility, particularly among older individuals. As the population of older PLWH continues to grow, co-occurring aging and HIV related declines in cognition and mobility will coincide; the effects of continued cannabis use In the Women's Interagency HIV Study (WIHS), it was found that current cannabis use was associated with over double the odds of single fall, and over 2.5 times the odds of multiple falls in 6 months; past cannabis use was associated with over 1.5 greater odds of single fall and multiple falls. Preliminary data shows that 40% of WIHS women (mean age 48) reported at least one fall over 2 years; current cannabis users had 1.7 times greater fall risk among HIV+ but not HIV-women. The hypothesis is that falls are related to acute effects of cannabis on attention and mobility, and that given subtle, pre-existing deficits associated with HIV infection, these acute cannabis effects may be more pronounced in HIV+ women, placing them at increased risks of falls. Whether this observed fall risk associated with cannabis use represents acute effects, or persistent effects of past cannabis use on cognition, balance, or mobility, or whether adverse effects of cannabis differ by HIV status merits further study in this aging population.

The "Walking While Talking" (WWT) test requires individuals to walk while performing a secondary attention-demanding task (dual task), has been used to assess the interactions between cognition and gait, and provides a framework for evaluating the effect of divided attention, a facet of executive functions, on mobility. Increased dual task costs measured using WWT may help unmask subtle and latent cognitive abnormalities before they become clinically apparent by increasing the complexity of the walking condition, and predict falls, frailty, disability, and mortality among older community-residing adults. Because both cannabis use and HIV have been implicated in impairments in attention and executive functions, the WWT may be a quick and simple mobility stress test to identify subtle cognitive and motor effects of acute cannabis administration as a function of HIV status.

The objective is to explore the mechanisms that underlie the increased fall risk associated with cannabis use. The effects of controlled administration of active (7.0% THC) and inactive (0.0%) cannabis in aging HIV+ women on stable HAART and HIV- controls enrolled on the WIHS will be compared. Endpoints will be balance, mobility, and cognition, including a cognitive-motor divided attention task (WWT). Specific aims and hypotheses are:

1. To determine the acute effects of cannabis on balance and mobility among older HIV+ and HIV- women. These test will be performed within subject comparisons of performance on balance and mobility tests at two supervised visits, with administration of placebo vs. active cannabis in counter-balanced order. The hypothesis is that HIV+ women will have greater impairment on balance and mobility, especially on complex walking conditions that demand attention, with administration of active cannabis than HIV- women
2. To determine the acute effects of cannabis on cognition among older HIV+ and HIV- women.HIV+ women will have greater impairment on cognitive testing, especially in attention, with administration of active cannabis than HIV- women.

ELIGIBILITY:
Inclusion Criteria:

1. current cannabis use (within 6 months) based on self-report
2. able to perform study procedures, including ability to ambulate independently
3. adequate hearing and vision
4. for HIV+ women use of stable HAART for at least 6 months.

Exclusion Criteria:

1. pregnancy
2. current illicit drug use other than cannabis
3. request for substance use treatment
4. current parole or probation
5. recent history of significant violent behavior (within 12 months)
6. major current Axis I psychopathology (e.g.,bipolar disorder, suicide risk, schizophrenia)
7. current use of psychiatric medication known to influence cognition
8. significant uncontrolled medical illness (such as uncontrolled diabetes or hypertension, clinically significant laboratory abnormalities, liver function tests (LFTs)>3x upper limit of normal)
9. history of active heart disease within 12 months
10. history of dementia
11. severe hand tremor
12. history of Central Nervous System (CNS) diseases or injury
13. poor English fluency.

All participants will be consented and compensated for their effort as approved by the Institutional Review Boards (IRBs) of each participating institution (see human subjects).

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only cohort
Enrollment: 25 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Sharma, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this study is an essential part of our proposed activities and will be carried out in terms of presentations at national and international scientific meetings as well as with publications in peer-reviewed journals. We would wish to make our results available to the community of scientists interested in understanding the consequences of substance use in older persons living with HIV, to foster future collaborative efforts and to avoid unintentional duplication of research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sets can be shared once analysis has been completed.
Access Criteria: The Data Analysis and Coordination Center (DACC) shares data to all investigators (internal and external) with Executive Committee (EC)-approved concept sheets. The concept sheet form requests information on the project background, specific aims and hypotheses, study design, laboratory and quality assurance methods, and plans for data analysis. All requests should be submitted online.
URL: https://statepi.jhsph.edu/mwccs/data-sharing/

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes: Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Placebo 0% THC cigarettes will be administered to HIV positive women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV positive women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes: Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Placebo 0% THC cigarettes will be administered to HIV negative women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV negative women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
  Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
Period: First Intervention (< 1 Day)
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Started | 10 | 4 | 5 | 6
Completed | 10 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Washout (From 1 Day to 212 Days)
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Started | 10 | 4 | 5 | 6
Completed | 8 | 3 | 5 | 5
Not Completed | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1
Period: Second Intervention (< 1 Day)
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Started | 8 | 3 | 5 | 5
Completed | 8 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants shown in their originally assigned study arm/group.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | Total
Number analyzed (Participants) | 10 | 4 | 5 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 5 | 6 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48.0 [46.0 to 54.0] | 56.5 [50.0 to 59.5] | 50.0 [42.0 to 51.0] | 45.5 [39.0 to 53.0] | 50 [44 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 5 | 6 | 25
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 4 | 5 | 16
  Not Hispanic or Latino | 5 | 2 | 1 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Due to small sample size Race data was stratified by "Black" vs "Non-Black"
  participants
    Non Black | 3 | 1 | 0 | 1 | 5
    Black | 7 | 3 | 5 | 5 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 | 5 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Acute Effects of Cannabis on Mobility Gait Speed (m/s)
Description: Mobility Gait Speed will be tested using the timed gait speed test. Gait speed is measured and reported under normal walking and attention demanding measures. Change in mobility as a function of timed gait speed from before cannabis, or placebo use, to after cannabis, or placebo, use at the 15 minute and 60 minute timepoints will be assessed. The baseline measurement, the mean of the two timepoint measurements, changes from the baselines, and change from the baseline to mean of 15 & 60 minutes for Cannabis minus that for Placebo, will be reported in meters/second (m/s).
Time Frame: Baseline, 15 minutes, and 60 minutes after taking cannabis or placebo during first visit. Duration between 1st and 2nd visits up to 7 months apart
Measure: Mean (Standard Error); unit: m/s
Groups:
- HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes; HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes: Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV positive women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV negative women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Number analyzed (Participants) | 8 | 3 | 5 | 5
m/s
  Baseline using Placebo | 2.89 (0.16) | 3.11 (0.54) | 2.87 (0.26) | 2.99 (0.32)
  Mean of 15 minute and 60 minute timepoint using Placebo | 2.86 (0.15) | 3.16 (0.53) | 3.04 (0.23) | 2.92 (0.20)
  Change from Baseline using Placebo | -0.03 (0.09) | 0.05 (0.19) | 0.16 (0.05) | -0.07 (0.14)
  Baseline using Cannabis | 2.80 (0.17) | 3.34 (0.70) | 2.59 (0.33) | 3.05 (0.31)
  Mean of 15 minute and 60 minute timepoint using Cannabis | 2.82 (0.12) | 3.03 (0.59) | 2.80 (0.34) | 3.14 (0.18)
  Change from Baseline using Cannabis | 0.02 (0.14) | -0.31 (0.25) | 0.21 (0.05) | 0.08 (0.20)
  Change from Baseline to Mean of 15 & 60 minutes for Cannabis minus that for Placebo | 0.05 (0.11) | -0.35 (0.45) | 0.04 (0.05) | 0.15 (0.14)
Statistical Analysis 1: Comparison: HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes vs HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes; Hypothesis Being Tested in 2 way ANOVA is that the difference in the change from Baseline to the Average of 15 and 60 minutes post baseline while on cannabis Vs. the change while on placebo (i.e. the last row in the outcomes) is greater for HIV+ subjects than for HIV- subjects; Test type: Superiority; p = 0.17, ANOVA

2. Primary Outcome: Change in Acute Effects of Cannabis on Balance - Functional Reach (cm)
Description: Change in balance from baseline will be tested using the Functional Reach test. Functional reach measures the distance the subject can reach in front of them from a standing position without losing balance. Change in balance from before cannabis, or placebo, use to after cannabis, or placebo, use at the 15 minute and 60 minute timepoints will be assessed. The baseline measurement, the mean of the two timepoint measurements, changes from the baselines, and change from the baseline to mean of 15 & 60 minutes for Cannabis minus that for Placebo, will be reported in centimeters (cm).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: cm
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Number analyzed (Participants) | 8 | 3 | 5 | 5
cm
  Baseline using Placebo | 28.22 (2.58) | 18.77 (3.36) | 36.75 (5.15) | 29.72 (3.74)
  Mean of 15 minute and 60 minute timepoint using Placebo | 26.92 (3.32) | 26.40 (5.72) | 32.13 (5.93) | 28.21 (3.95)
  Change from Baseline using Placebo | -1.30 (1.66) | 3.64 (2.84) | -4.61 (1.63) | -1.51 (0.79)
  Baseline using Cannabis | 28.71 (3.71) | 22.39 (4.59) | 31.34 (3.82) | 34.26 (6.06)
  Mean of 15 minute and 60 minute timepoint using Cannabis | 29.65 (4.00) | 18.04 (3.09) | 33.87 (4.51) | 30.93 (2.37)
  Change from Baseline using Cannabis | 0.94 (3.71) | -4.35 (2.36) | 2.52 (1.60) | -3.33 (3.98)
  Change from Baseline to Mean of 15 & 60 minutes for Cannabis minus that for Placebo | 2.24 (3.41) | -7.99 (3.79) | 7.14 (2.01) | -1.82 (4.64)
Statistical Analysis 1: Comparison: HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes vs HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.18, ANOVA

3. Primary Outcome: Change in Acute Effects of Cannabis on Cognition Using Sustained Attention Response Test (% Correct Suppressions)
Description: Cognition will be tested using the number of correct suppressions on the Sustained Attention to Response Task (SART). Participants were asked to respond to a series of digits on a computer screen by pressing a key as quickly as possible for every digit except "3". The percentage of correct suppressions is quantified. Change in the percentage of mean correct suppressions before cannabis (or placebo) use to after cannabis (or placebo) at the 15 minute and 60 minute timepoints will be assessed. The baseline measurement, the mean percentage of the two timepoint measurements, the mean percentage changes from baseline values, and change from the baseline to mean of 15 & 60 minutes for Cannabis minus that for Placebo, will be reported.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of correct suppressions
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes
Number analyzed (Participants) | 8 | 3 | 5 | 5
Percentage of correct suppressions
  Baseline using Placebo | 84.00 (1.51) | 64.00 (16.17) | 87.40 (3.71) | 79.20 (9.75)
  Mean of 15 minute and 60 minute timepoint using Placebo | 82.25 (2.25) | 78.67 (6.77) | 74.00 (10.62) | 78.40 (10.05)
  Change from Baseline using Placebo | -1.75 (2.25) | 14.67 (10.09) | -12.40 (8.01) | -0.80 (7.58)
  Baseline using Cannabis | 80.50 (5.58) | 85.33 (2.67) | 90.40 (4.49) | 80.00 (12.77)
  Mean of 15 minute and 60 minute timepoint using Cannabis | 85.50 (2.80) | 88.67 (3.53) | 80.00 (7.80) | 78.00 (13.90)
  Change from Baseline using Cannabis | 5.00 (3.96) | 3.33 (1.33) | -10.00 (8.01) | -2.00 (1.67)
  Change from Baseline to Mean of 15 & 60 minutes for Cannabis minus that for Placebo | 6.75 (5.14) | -11.33 (11.10) | 2.00 (5.10) | -1.20 (9.02)
Statistical Analysis 1: Comparison: HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Positive: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes vs HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes First, Then Placebo 0% THC Cigarettes vs HIV Sero Negative: Placebo 0% THC Cigarettes First, Then Cannabis 7% delta9-THC Cigarettes; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.72, ANOVA

ADVERSE EVENTS:
Time Frame: Participants were monitored during the two study visits, up to approximately 7 months total
Groups:
- HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes; HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes: Drug: Cannabis 7% delta9-THC cigarettes will be smoked by 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Positive: Placebo 0% THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV positive women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
- HIV Sero Negative: Placebo 0% THC Cigarettes: Placebo 0% THC cigarettes will be administered to HIV negative women. Participants will be instructed to 'light the cigarette' (30 sec), 'get ready' (5 sec), 'inhale' (5 sec), 'hold smoke in lungs' (10 sec) and 'exhale.' Participants will smoke 3 puffs in this manner, with a 40-sec interval between each puff.
Arm/Group | HIV Sero Positive: Cannabis 7% delta9-THC Cigarettes | HIV Sero Positive: Placebo 0% THC Cigarettes | HIV Sero Negative: Cannabis 7% delta9-THC Cigarettes | HIV Sero Negative: Placebo 0% THC Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT03633721/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03633721/ICF_001.pdf